CLINICAL TRIAL: NCT00035620
Title: A Study of Single Dose Per Cycle Filgrastim-SD/01 as an Adjunct to VAdriaC/IE Chemotherapy in Pediatric Sarcoma Patients
Brief Title: Pegfilgrastim as Support to Pediatric Sarcoma Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 990130
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Sarcoma; Neutropenia
Keywords: Bone cancer; Sarcoma; Neutropenia; Chemotherapy
MeSH Terms: conditions — Sarcoma; Neutropenia; Bone Neoplasms | interventions — pegfilgrastim; Filgrastim

ARMS (2):
- Filgrastim (Active Comparator): Filgrastim
  Interventions: Drug: filgrastim
- Pegfilgrastim (Experimental): Pegfilgrastim
  Interventions: Drug: pegfilgrastim

INTERVENTIONS:
Drug: pegfilgrastim — pegfilgrastim
  Arms: Pegfilgrastim
Drug: filgrastim — filgrastim
  Arms: Filgrastim

SUMMARY:
Physicians are conducting a clinical trial for patients with pediatric sarcoma. Sarcoma is a type of bone cancer that can be treated with chemotherapy which can affect the bone marrow, where blood cells are produced. Neutrophils are a type of white blood cells that fight infection and are produced in the bone marrow. If the neutrophil count becomes too low due to chemotherapy, a potentially serious condition called neutropenia occurs. Neutropenia is serious because it can affect the body's ability to protect against many types of infections. Pegfilgrastim is an investigational drug being evaluated for its potential ability to increase the number of neutrophils. The purpose of this study is to determine the safety and effectiveness of pegfilgrastim in preventing neutropenia following chemotherapy in pediatric patients up through the age of 21 with sarcoma.

ELIGIBILITY:
* Sarcoma * No previous chemotherapy or radiotherapy * Patients who will be receiving chemotherapy consisting of Vincristine, Doxorubicin, Cyclophosphamide, Etoposide, Ifosfamide, and Mesna

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2000-04; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Duration of severe neutropenia in chemotherapy in cycles 1 and 3 | cycles 1 and 3
Time to ANC recovery to greater than or equal to 0.5 x 10^9/L in cycles 1 and 3 | cycles 1 and 3

SECONDARY OUTCOMES:
Pharmacokinetic profile in chemotherapy cycles 1 and 3 | cycles 1 and 3
Incidence of adverse events across all cycles of chemotherapy | all cycles
Overall rates of febrile neutropenia | all cycles

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_990130.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/